CLINICAL TRIAL: NCT00274274
Title: Efficacy and Safety of Insulin Aspart in a Fixed or Flexible Supplementary Insulin Therapy Regimen, With or Without Insulin Detemir in Type 2 Diabetes
Brief Title: Efficacy and Safety of a Fixed or a Flexible Supplementary Insulin Therapy in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1657; 2005-000319-87 (EudraCT Number)
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe. This trial aims for a comparison of the efficacy and safety of Insulin Aspart, given in a fixed or in a flexible supplementary insulin therapy, with or without Insulin Detemir plus Metformin, if needed, in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes for more than 6 months
* Treatment with 1 or more oral anti-diabetic drugs or insulin, or a combination of these for more than 3 months
* Body Mass Index (BMI) less than or equal to 40 kg/m2
* HbA1c 7.0-11.0%

Exclusion Criteria:

* Treatment with short acting insulin(s) for longer than 10 days
* Current treatment with TZDs. A TZD medication must be stopped at least 14 days before the randomization
* Proliferative retinopathy or maculopathy requiring acute or laser treatment within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2005-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 52 weeks

SECONDARY OUTCOMES:
Blood glucose profiles
Percentage of patients with HbA1c less than 7.0% after 52 weeks
Quality of Life
Frequency of BG measurements
Safety parameters
Duration of education

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Düsseldorf, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com